CLINICAL TRIAL: NCT00852878
Title: The Treatment of Recurrent Abdominal Pain in Children: A Comparison of Biofeedback and Behavioral Intervention
Brief Title: The Treatment of Recurrent Abdominal Pain in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough interested participants
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPSC IRB #5275
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2010-12

CONDITIONS: Recurrent Abdominal Pain
Keywords: Recurrent Abdominal Pain; Biofeedback; Heart Rate Variability
MeSH Terms: conditions — Abdominal Pain | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biofeedback (Active Comparator): heart rate variability biofeedback
  Interventions: Behavioral: Biofeedback
- Behavioral (Active Comparator): Behavioral intervention will provide parent and child with a variety of pain management techniques such as relaxation, distraction, contingency management, and coping statements
  Interventions: Behavioral: Behavioral Protocol

INTERVENTIONS:
Behavioral: Biofeedback — Biofeedback will teach resonant frequency breathing for 6-8 sessions
  Other Names: resonant frequency breathing
  Arms: Biofeedback
Behavioral: Behavioral Protocol — Behavioral protocol will teach a variety of pain management techniques such as relaxation, distraction, and coping statements over 6-8 sessions
  Other Names: relaxation, distraction, and coping statements
  Arms: Behavioral

SUMMARY:
The purpose of this study is to determine if two treatments, a biofeedback and behavioral protocol, for recurrent abdominal pain are equally effective.

DETAILED DESCRIPTION:
Recurrent abdominal pain (RAP) is a functional disorder that affects approximately 10 to 25% of children in the United States. This population tends to be heavy medical users in a search of a treatment for the chronic pain, but at this time there is no standard treatment protocol. The literature proposes that there are two effective treatments for RAP, a relaxation protocol by Sanders et al. (1994) and a biofeedback protocol currently in use at Kaiser, but neither treatment has been widely accepted as standard treatment. A purpose of this study is to gather more data on both treatments to help move one or both treatments into the standard of care for RAP. The hypothesis of this study is that the biofeedback and the relaxation protocols will have equivalent treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* who speak English
* diagnosis with Recurrent abdominal pain

Exclusion Criteria:

* lactose intolerance, urinary tract infections, or recent head trauma;
* the use of prescribed or over he counter medications, which may interfere with the biofeedback data;
* currently receiving other treatment for recurrent abdominal pain;
* the receipt of a recent and related surgical procedure;
* children who met criteria for depression or anxiety disorder

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
The measurable primary outcome will use equivalency testing on changes in pain diary ratings, using the average weekly pain intensity and frequency as recorded in the pain dairy | 3 Months

SECONDARY OUTCOMES:
A measurable secondary outcome will be changes in heart rate variability | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Warren L Shapiro, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Vandever Medical Offices, San Diego, California, United States